CLINICAL TRIAL: NCT03473288
Title: Rejuvenation of Aged Muscle Stem Cells Through Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment due to COVID restrictions and funding issues
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00084763; 1K01AG056664 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Autophagy and Apoptosis in Human Satellite Cells
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Treadmill Exercise (Active Comparator): Moderate intensity treadmill exercise three times per week for 10-12 weeks
  Interventions: Behavioral: Exercise
- Sedentary Controls (Placebo Comparator): Serve as a sedentary (little exercise) control for 10-12 weeks
  Interventions: Behavioral: Sedentary

INTERVENTIONS:
Behavioral: Exercise — Participants will undergo supervised exercise 3 times a week for 10-12 weeks.
  Arms: Moderate Intensity Treadmill Exercise
Behavioral: Sedentary — Participants will be asked to maintain the sedentary lifestyle that they already have for 10-12 weeks.
  Arms: Sedentary Controls

SUMMARY:
The proposed study will establish a newly-identified signaling pathway regulating both autophagy and apoptosis in human satellite cells. These findings will allow for novel pharmacological targets in satellite cells to return regenerative capacity to elderly individuals. Up to 80 adults, 21 years of age and greater, will undergo a consent visit followed by three blood draws and muscle biopsy visits- baseline (pre), after the first exercise bout (post-acute), and after the 12 week training program (post-chronic). Blood will be obtained and tested for inflammatory (IL-6/TNF/IL-1) and endocrine markers (Testosterone/Estrogen/Thyroid hormone). As part of the intervention, participants will undergo moderate intensity treadmill exercise three times per week for 10-12 weeks or serve as sedentary controls. Muscle stem cell function will be compared across age groups at each time point using a One Way ANOVA or t test for specific comparisons. An alternative analysis will be a longitudinal design following muscle stem cell function from each individual before and after exercise training. This analysis will be performed with repeated measure ANOVAs. Data will be analyzed using GraphPad Prism 6 statistical software. Significance will be accepted as p<.05. Thigh Muscle biopsies may result in momentary pain and discomfort, burning or bleeding, numbness, and rarely fainting or infection. The incision site may leave a scar and muscle soreness may be present up to ten days after the biopsy. While the local numbing medicine xylocaine is almost entirely free from allergic properties (such as causing hives), an allergic reaction is possible, and the participant will not be given xylocaine if they have a history of such a reaction. The xylocaine will be given by a small injection into the skin at the site of the muscle biopsy. Risks associated with a standard blood draw include momentary discomfort and/or bruising. In addition, there is a minimal risk of infection, excess bleeding, clotting, and fainting. An exercise program may result in muscle, bone and/or joint soreness, discomfort and/or injury. All collected data will be stored in a locked file to be accessed only by Dr. White and his study staff. Study records that identify subjects will be kept confidential as required by law.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or greater.
* No medication changes within the last 3 months.
* Not participating in regular physical exercise (more than 60 minutes of moderate intensity or 30 minutes of vigorous intensity exercise per week).
* Able to decide if you want to take part in the study.

Exclusion Criteria:

* Smoker: Tobacco use within the last 12 months.
* Dieting or intending to diet.
* Use of potential confounding medications, e.g. using ticlopidine, clopidogrel, dipyridamole, warfarin, heparin, enoxaparin and other blood thinners.
* Coronary stents or any other medical condition for which aspirin cannot be temporarily withheld.
* Use of hormone replacement medications.
* Absolute contra-indications to exercise: Recent (<6 months) acute cardiac event unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurysm and acute systemic infection.
* Relative contra-indications to exercise: Left main coronary stenosis, moderate stenotic valvular heart disease, outflow tract obstruction, high degree AV block, ventricular aneurysm, uncontrolled metabolic disease (e.g. diabetes, thyrotoxicosis, myxedema), uncontrolled pulmonary disease (e.g. severe COPD or pulmonary fibrosis), mental or physical impairment leading to inability to exercise adequately.
* Have a confounding medical condition that is progressive and unstable such as HIV, Hepatitis C, active cancer, and/or taking medications for those conditions.
* Unwillingness to be randomized to any one of two intervention groups, submit to skeletal muscle biopsies and all other study testing or continuously participate in a randomly assigned exercise training or program for three months.
* Orthopedic limitations, musculoskeletal disease and/or injury.
* Allergic to xylocaine.
* Unwillingness to exercise at the Duke Center for Living during staff supervised times.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Stem Cell Function by Age Group | Baseline, 1 Week Post Baseline, and 12 Weeks Post Baseline
  Muscle stem cell function will be compared across age groups at baseline, post-acute (1 week after baseline), and post-chronic (12 weeks after baseline) using a One Way ANOVA or t test for specific comparisons

CONTACTS AND LOCATIONS:
Overall Officials: James White, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03473288/Prot_000.pdf